CLINICAL TRIAL: NCT04457466
Title: Assessment of the Effects of Extensive Sensorimotor Training on Pain Processing
Brief Title: Assessment of the Effects of Extensive Somatosensory Training on Pain Processing
Status: Terminated | Type: Observational
Why Stopped: Covid-19
Sponsor: Aalborg University (Other)
Collaborators: University of Aarhus (Other); Lundbeck Foundation (Other); Danish National Research Foundation (Other)
Responsible Party: Principal Investigator, Anna M. Zamorano, Principal Investigator, Aalborg University
Other Study IDs: 10042017
Record Dates: First submitted 2020-06-24; First posted 2020-07-07 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Nerve Growth Factor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy musicians: Men and women aged 18-60, who must be enrolled in a music conservatory performance program or be professionally active, and must speak and understand English.
  Interventions: Drug: Nerve Growth Factor
- Healthy non-musicians: Men and women aged 18-60, must speak and understand English and not have any kind of musical training.
  Interventions: Drug: Nerve Growth Factor
- Musicians with chronic pain: Men and women aged 18-60 with chronic and idiopathic musculoskeletal upper limb and/or neck pain lasting more than 6 months. They must be enrolled in a music conservatory performance program or be professionally active and must speak and understand English.
  Interventions: Drug: Nerve Growth Factor
- Non-musicians with chronic pain: Men and women aged 18-60 with chronic and idiopathic musculoskeletal upper limb and/or neck pain lasting more than 6 months. They must not have any kind of musical training and must speak and understand English.
  Interventions: Drug: Nerve Growth Factor

INTERVENTIONS:
Drug: Nerve Growth Factor — Induction of experimental muscle soreness using intramuscular injections of Nerve Growth Factor.

SUMMARY:
Persistent pain may lead to several alterations in the brain activity and sensory perception (i.e. pain). Around 80% of professional musicians experience prolonged episodes of musculoskeletal pain throughout their careers, a percentage that is four times higher than in the general population. With this background, the intended experiment aims at understanding the role of several biological factors associated to sensorimotor training that can lead to alteration of the brain activity and, consequently, pain processing.

ELIGIBILITY:
Inclusion Criteria:

Healthy men and women Speak and understand English.

General exclusion criteria are:

* Pregnancy
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Previous neurologic or mental illnesses
* Presence of a history of trauma or neurologic entrapment syndromes to the arm regions.
* Lack of ability to cooperate
* Frequent computer gamer ( > 9 hours/week)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy men and women Speak and understand English.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Pain rating | Changes from baseline measured at day 3 and day 8
  Pain on an 11-point numerical rating scale (0 = no pain, 10 = most intense pain imaginable)
Cortical Sensory Evoked Potentials | Changes from baseline measured at day 3 and day 8
  Electrical stimulation will be elicited to record sensory evoked potentials using electroencephalography (EEG)
Motor Evoked Potentials | Changes from baseline measured at day 3 and day 8
  Transcranial magnetic stimualtion will be used to evoke motor evoked potentials (MEPs)
Brain connectivity | Changes from baseline measured at day 3 and day 8
  Continuous electroencephalography recording will be used to explore connectivity between brain areas

SECONDARY OUTCOMES:
Questionnaires | Changes from baseline measured at day 3 and day 8
  Questionnaires about pain and muscle soreness (Pain catastrophization; State and Trait anxiety; Pain vigilance)
Pressure pain thresholds | Changes from baseline measured at day 3 and day 8
  Pressure applied to the surface of the skin using a handheld algometer

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zamorano AM, Kleber B, De Martino E, Insausti-Delgado A, Vuust P, Flor H, Graven-Nielsen T. Prior use-dependent plasticity triggers different individual corticomotor responses during persistent musculoskeletal pain. Pain. 2025 Jul 30. doi: 10.1097/j.pain.0000000000003749. Online ahead of print. PMID 40728516